CLINICAL TRIAL: NCT01872208
Title: A Pilot Study for Evaluation of the Safety and Efficacy of Humacyte's Human Acellular Vascular Graft as an Above-Knee Femoro-Popliteal Bypass Graft in Patients With Peripheral Arterial Disease
Brief Title: Evaluation of the Safety and Efficacy of a Vascular Prosthesis as an Above-Knee Bypass Graft in Patients With PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V002
Record Dates: First submitted 2013-05-22; First posted 2013-06-07 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease
Keywords: PAD; Atherosclerosis; Peripheral circulation; Blood Vessel Prosthesis; Tissue-Engineered Vascular Graft; Vascular Prosthesis Implantation; Femoro-Popliteal Bypass
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Human Acellular Vessel (HAV) (Experimental): HAV implantation to study participants.
  Interventions: Biological: HAV implantation

INTERVENTIONS:
Biological: HAV implantation — Patients will be implanted with a Human Acellular Vessel (HAV) as an above-knee femoro-popliteal bypass graft using standard vascular surgical techniques.
  Other Names: Human Acellular Vessel

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a novel, tissue-engineered vascular prosthesis, the Human Acellular Vessel (HAV).

The HAV is intended as an alternative to synthetic materials and to autologous grafts in the creation of an above-knee femoro-popliteal bypass graft in patients with peripheral arterial disease.

DETAILED DESCRIPTION:
The HAV is a sterile, non-pyrogenic, acellular tubular graft composed of human collagens and other natural extra-cellular matrix proteins. Upon implantation, it is anticipated (based on pre-clinical studies) that the collagen-based matrix comprising the graft will be infiltrated with host cells and re-modeled by the host. This will result in a vascular structure more similar to the histological composition of the native vascular tissue that may improve graft longevity and be less likely to become infected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic peripheral arterial disease who require above knee femoro-popliteal bypass surgery
* Claudication distance of 200 m or less or rest pain or critical limb ischemia
* Preoperative angiography or angio-CT shows superficial femoral artery occlusion of >10 cm AND graft length required ≤ 30 cm. This imaging may have been conducted up to 3 months prior to study entry provided that the patient's symptoms have remained stable since that time
* Preoperative imaging shows at least two below knee vessels patent to the ankle with good runoff
* Femoral artery occlusion is not considered suitable for endovascular treatment
* Autologous vein grafts are not suitable or feasible e.g. because of severe venous disease or prior use of leg veins for other bypass surgery or there is a clinical need to preserve those veins for future bypass surgery in the coronary or peripheral circulation
* Aged 18 to 80 years old, inclusive
* Hemoglobin ≥ 10 g/dL and platelet count ≥ 100,000/mm3 prior to Day 1
* Other hematological and biochemical parameters within a range considered acceptable for the administration of general anesthesia prior to Day 1
* Adequate liver function, defined as serum bilirubin ≤ 1.5 mg/dL; GGT, AST, ALT, and alkaline phosphatase ≤ 2x upper limit of normal or INR ≤ 1.5 prior to Day 1.
* Able to communicate meaningfully with investigative staff, competent to give written informed consent, and able to comply with entire study procedures
* Able and willing to give informed consent
* Life expectancy of at least 2 years

Exclusion Criteria:

* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months prior to study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* Acute injury or active infection (including positive cultures of pathogenic bacteria) in the limb receiving the graft
* Stroke within six (6) months prior to study entry (Day 1)
* Treatment with any investigational drug or device within 60 days prior to study entry (Day 1)
* Women of child bearing potential
* Active diagnosis of cancer within the previous year
* Immunodeficiency including AIDS / HIV
* Documented hypercoagulable state or history of 2 or more DVTs or other spontaneous intravascular thrombotic events
* Bleeding diathesis
* Ongoing treatment with vitamin K antagonists or direct thrombin inhibitors or factor Xa inhibitors (e.g. dabigatran, apixaban or rivaroxaban)
* Previous arterial bypass surgery (autologous vein or synthetic graft) in the operative limb
* Previous angioplasty with stenting in the operative limb unless the graft anastomoses can be made at least 1cm distant from the site of the stent
* Stenosis of >50% of the external iliac artery unless it is planned to treat this stenosis with angioplasty with or without stenting prior to, or at the time of, graft implantation
* Distal graft anastomosis likely to be below the knee
* Active autoimmune disease - symptomatic or requiring ongoing drug therapy
* Active local or systemic infection (WBC > 15,000/mm3)
* Known serious allergy to aspirin or penicillin
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the HAVG
* Previous enrollment in this study
* Employees of the sponsor or patients who are employees or relatives of the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-10-10 (Actual); Primary Completion 2016-05-30 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Change in HAV characteristics | From day 5 to month 24 after HAV implantation.
  The incidence of aneurysm formation, anastomotic bleeding or rupture, graft infection and irritation/inflammation/infection at the implantation site will be assessed by Doppler ultrasound and tabulated.
Change in HAV patency rate | From day 5 to month 24 after HAV implantation.
  Determine the patency (primary, primary assisted and secondary) rate of the Humacyte HAV by Doppler ultrasound.
Change in frequency and severity of Adverse Events | From day 1 to month 24 after HAV implantation.
  Frequency and severity of AEs of each patient will be documented.
Change in hematology, coagulation and clinical chemistry parameters | From baseline to week 26 after HAV implantation.
  Change from baseline in hematology, coagulation and clinical chemistry parameters.

SECONDARY OUTCOMES:
Change from baseline in Panel Reactive Antibody (PRA) | From baseline to week 26 after HAV implantation.
  Assess changes in the Panel Reactive Antibody response over 6 months after graft implantation.
Development of IgG antibodies | From baseline to week 26 after HAV implantation.
  Determine whether IgG antibodies to the extracellular matrix material are formed in response to implantation of the HAVG over the 6 months after implantation.
HAV patency rates | At months 6, 12, 18 after HAV implantation.
  To determine the patency rates of the graft (primary, primary assisted and secondary).
Graft interventions | At days 5, 15, weeks 6, 12, 16, months 12, 18, 24 after HAV implantation.
  Determine the rates of interventions needed to maintain / restore patency in the graft.
Effect of graft implantation on PAD symptoms | From baseline to weeks 6, 12, 26, months 12, 18, 24 after HAV implantation.
  Assessment of any effect of graft implantation on claudication, rest pain and ischemic ulcers.
Effect of graft on ankle-brachial index (ABI) | From baseline to weeks 6, 12, 26, months 12, 18, 24 after HAV implantation.
  Assessment of any effect of the graft on ankle-brachial index (ABI).

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, MD, Study Director — Humacyte, Inc.
Locations (3):
- Poland (3):
  - Clinic of Vascular Surgery and Angiology; Medical University in Lublin, Lublin
  - Pomeranian University in Szczecin; Clinic of General, Vascular Surgery and Angiology, Szczecin
  - Regional Specialist Hospital in Wroclaw; Clinic of Vascular Surgery, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gutowski P, Gage SM, Guziewicz M, Ilzecki M, Kazimierczak A, Kirkton RD, Niklason LE, Pilgrim A, Prichard HL, Przywara S, Samad R, Tente B, Turek J, Witkiewicz W, Zapotoczny N, Zubilewicz T, Lawson JH. Arterial reconstruction with human bioengineered acellular blood vessels in patients with peripheral arterial disease. J Vasc Surg. 2020 Oct;72(4):1247-1258. doi: 10.1016/j.jvs.2019.11.056. Epub 2020 Feb 21. PMID 32093913
- See also: Results of the clinical study have been published — http://pubmed.ncbi.nlm.nih.gov/32093913/